CLINICAL TRIAL: NCT03535181
Title: Pulsatility Aneurysmal Evaluation Process by Cerebral Dynamic CTA (Computed Tomography Angiography)
Acronym: PULSAN
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PULSAN (29BRC18.0073)
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-01

CONDITIONS: Aneurysm, 4D CT Scan
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intracranial aneurysm are frequent with a prevalence estimated over 2-5% in the general population. These are focal dilatations occuring in the cerebral vessels. They usually remain silent until complications occur. Complications associated with intracranial aneurysms include mass effect on adjacent structures and rupture. Rupture is the most severe complication with a mortality rate of 35-50% and a high rate of morbidity including long-term disability. It incidence is estimated about 1% per year for aneurysm smaller than 1 cm.

However, preventative treatments have their own risk of complication and morbi-mortality rate including stroke and hemorrhage. Actual guidelines for treatment planning are mainly designed with the size, the location and the age of the patient. This is why working on the identification of imaging markers of aneurysmal instability is relevant.

Dynamic CTA (Computed Tomography Angiography) acquisition allow to study the variation of metrics such as dome height, dome length, ostium width, ostium area, and volume during the cardiac cycle. The goal of this study is to assess different aneurysmal metrics to determine those which may vary the most during the cardiac cycle and to assess it as an imaging marker of aneurysmal instability.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an intracranial aneurysm assessed with a 4D CTA

Exclusion Criteria:

* Minor
* Refusal to participate

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients suffering from at least one intracranial aneurysm and who benefited from a 4D CTA in our institution.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Assess the variation of different aneurysmal metrics (dome height, dome length, ostium width, ostium area, and volume) during the cardiac cycle. | 6months
  Is there a difference between the maximum and the minimum values ? Measurements are realised with a 4D computed tomography angiography.

SECONDARY OUTCOMES:
Evaluate among different aneurysmal metrics (dome height, dome length, ostium width, ostium area, and volume) the most relevant ones. | 6months
  Evaluate among different aneurysmal metrics (dome height, dome length, ostium width, ostium area, and volume) for a composite endpoint including those which may vary the most during the cardiac cycle (maximum minus minium values) and which have the best reproducibilities over one (intrareader agreement) and multiples cardiac cycles.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France